CLINICAL TRIAL: NCT01509976
Title: Triclosan, Triclocarban, and the Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Julie Parsonnet, Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: AVOCET
Record Dates: First submitted 2012-01-06; First posted 2012-01-13 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Triclosan Effects on Microbial Flora
Keywords: Triclosan; Triclocarban; Microbial flora; Obesity
MeSH Terms: conditions — Obesity | interventions — Triclosan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Red (Other): This arm will either start with personal care products that contain triclosan and then and cross over to personal care products that do not contain triclosan or vice-versa. Since the investigators are blinded, it is not clear which arm is which.
  Interventions: Other: triclosan/triclocarban-containing personal care products
- Blue (Other): This arm will either start with personal care products that contain triclosan and then and cross over to personal care products that do not contain triclosan or vice-versa. Since the investigators are blinded, it is not clear which arm is which.
  Interventions: Other: triclosan/triclocarban-containing personal care products

INTERVENTIONS:
Other: triclosan/triclocarban-containing personal care products — Subjects will be randomly assigned to one of two arms with either triclosan/triclocarban-containing personal care products or products without triclosan/triclocarban. After 5 months, each subject will cross over to the other arm.

SUMMARY:
Triclosan (5-chloro-2 (22,4-dichlorophenoxy)phenol) is a broad-spectrum antibacterial and antifungal agent that is found in thousands of common household products, including deodorants, toothpaste, "antibacterial" soaps, cleaning products, kitchen utensils, bedding, socks, trash bags. The benefits of triclosan have not been proven except in reducing plaque and gingivitis when used in toothpaste. In this study, the investigators intend to look at whether exposure to triclosan changes the colonizing flora of the skin, gut and mouth as well as changes in certain blood hormone levels, including adipocytokines, androgens, and inflammatory markers. Changes in the gut microbiota have been associated with a variety of disease states such as inflammatory bowel disease, colorectal cancer. Additionally, reductions in the microbiome diversity have been associated with obesity.

DETAILED DESCRIPTION:
Hypothesis: Exposure to triclosan changes microbial flora and leads to changes in

Objectives:

1. Assess diversity and quantities of microbial flora in gut, skin, mouth before, during, and after TC use
2. Assess whether TC use correlates with microbial resistance
3. If any, assess time to change in alterations in microbial flora

Study design:

Prospective, randomized, double-blinded, cross-over study of 20 subjects

Here, we propose a pilot study in which we will compare the microbial flora of subjects who use triclosan-containing personal hygiene products and those who use triclosan-free products. We will randomize half the cohort to triclosan-containing personal hygiene products including toothpaste, liquid hand soap, bar soap, and dish soap for half of the cohort for a 5-month period of time. The participants and investigators will be blinded as to whether they are using triclosan-containing products or triclosan-free products by blinding the packaging. After about 5 months, the participants will cross-over to the other arm.

During a lead-in period of about 2 weeks, we will collect urine samples for a baseline triclosan level and body weight. We will also collect Leptin, Resistin, Grehlin, IL 10, IL17, PAI-1 Plasminogen activator inhibitor -1, TNFa, IFN-g, Insulin, IGF, Glucagon, CRP, TSH, Free T4T3, Estradiol, Testosterone free, Testosterone total, Adiponectin, IL6, Visfatin, H. pylori, ESR. Blood, urine, and body weight will be collected at three points in the study: prior to first phase, in between phases, and after completion of second phase.

We will collect stool, skin, tooth, and saliva samples multiple times throughout the study and submit for pyrosequencing.

ELIGIBILITY:
Inclusion Criteria:

* Health subjects
* Age >18 years

Exclusion Criteria:

* Pregnancy
* Recent travel to the developing world (within 3 months)
* Recent use of antibiotics (within 3 months)
* Unwillingness to change personal care/hygiene products
* Recent gastrointestinal illness (within 3 months)
* Individuals who are unlikely to be available for the 10 months of the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-07-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in microbial flora | 5 months in each phase for a total of 10 month study period
  We will assess diversity and quantities of microbial flora in gut, skin, mouth before, during, and after triclosan use.
Microbial resistance | 5 months in each phase for a total of 10 month study period
  We will assess whether triclosan use correlates with microbial resistance
Time to alteration in flora. | 5 months in each phase for a total of 10 month study period
  We will assess time to change in alterations in microbial flora, if any.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

REFERENCES:
- [Background] Turnbaugh PJ, Hamady M, Yatsunenko T, Cantarel BL, Duncan A, Ley RE, Sogin ML, Jones WJ, Roe BA, Affourtit JP, Egholm M, Henrissat B, Heath AC, Knight R, Gordon JI. A core gut microbiome in obese and lean twins. Nature. 2009 Jan 22;457(7228):480-4. doi: 10.1038/nature07540. Epub 2008 Nov 30. PMID 19043404
- [Background] Russell AD. Whither triclosan? J Antimicrob Chemother. 2004 May;53(5):693-5. doi: 10.1093/jac/dkh171. Epub 2004 Apr 8. PMID 15073159
- [Background] Queckenberg C, Meins J, Wachall B, Doroshyenko O, Tomalik-Scharte D, Bastian B, Abdel-Tawab M, Fuhr U. Absorption, pharmacokinetics, and safety of triclosan after dermal administration. Antimicrob Agents Chemother. 2010 Jan;54(1):570-2. doi: 10.1128/AAC.00615-09. Epub 2009 Oct 12. PMID 19822703
- [Background] Guyer B, Freedman MA, Strobino DM, Sondik EJ. Annual summary of vital statistics: trends in the health of Americans during the 20th century. Pediatrics. 2000 Dec;106(6):1307-17. doi: 10.1542/peds.106.6.1307. PMID 11099582
- [Background] Cummings DE, Schwartz MW. Genetics and pathophysiology of human obesity. Annu Rev Med. 2003;54:453-71. doi: 10.1146/annurev.med.54.101601.152403. Epub 2001 Dec 3. PMID 12414915
- [Background] Charles J, Pan Y, Britt H. Trends in childhood illness and treatment in Australian general practice, 1971-2001. Med J Aust. 2004 Mar 1;180(5):216-9. doi: 10.5694/j.1326-5377.2004.tb05888.x. PMID 14984340
- [Background] Strachan DP. Hay fever, hygiene, and household size. BMJ. 1989 Nov 18;299(6710):1259-60. doi: 10.1136/bmj.299.6710.1259. No abstract available. PMID 2513902